CLINICAL TRIAL: NCT03186040
Title: Open-label Clinical Trial: Safety of Lacosamide in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Open-label Clinical Trial of Lacosamide in ALS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Satoshi Kuwabara, Professor, Chiba University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G29007
Record Dates: First submitted 2017-06-05; First posted 2017-06-14 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Lacosamide

STUDY DESIGN:
Intervention Model Description: Before and after comparison
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lacosamide (Other)
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Sodium channel blocker

SUMMARY:
Lacosamide is administered for patients with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
Lacosamide is administered for patients with amyotrophic lateral sclerosis (ALS). This clinical trial is open-label, single group and before and after comparison study. Dosage of lacosamide is increased from 100mg to 400mg for 4 weeks. Safety of lacosamide administration in ALS is primary endpoint. Nerve excitability, fasciculation and muscle cramp are investigated before and after administration for secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 year old
* Probable or definite ALS disease evaluated by Awaji electrophysiological criteria
* Subjects provided informed consent.

Exclusion Criteria:

* Patient without ability to comprehend informed consent
* Patient with uncompensated medical illness
* Patient with cardiac disease (myocardial infarction, valvular disease and cardiomyopathy etc.)
* Patient with arrhythmia (incomplete atrioventricular block and bundle branch block etc.)
* Patient with sodium channel disorders, such as Brugada syndrome
* Patient already administered anti-arrhythmic drug which prolongs PR interval (interval between arterial and ventral contraction measured by ECG)
* Pregnant or breast-feeding woman
* Patient with forced vital capacity of < 60% predicted
* Patient already performed tracheotomy or tube feeding
* Patient who takes any other experimental agents 3 months before.
* Not enough compound muscle action potential amplitude in the median nerve to be performed nerve excitability test
* Patient who plans to change medicine which affects nerve excitability during this trial 4 weeks
* Familial ALS
* Patient who is judged inappropriate for this trail by doctors responsible for this trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | 4 weeks
  Adverse events will be observed at each visit by direct questioning of the subjects, clinical examination, electrocardiogram (ECG), vital signs, vital capacity and laboratory test results.

SECONDARY OUTCOMES:
Frequency of fasciculation | Baseline, Week 2 and Week 4
  Frequency of fasciculation measured by ultrasound and surface electromyogram at baseline, week 2 and week 4.
Frequency and extent of muscle cramp | Baseline, Week 2 and Week 4
  Frequency of muscle cramp and the extent of muscle cramp measured by visual analog scale (VAS) at baseline, week 2 and week 4.
Effects on strength-duration time constant | Baseline, Week 2 and Week 4
  Measured by threshold tracking nerve conduction studies
Effects on 0.2ms threshold change | Baseline, Week 2 and Week 4
  Measured by latent addition method
Effects on threshold electrotonus | Baseline, Week 2 and Week 4
  Measured by threshold tracking nerve conduction studies
Effects on recovery cycle | Baseline, Week 2 and Week 4
  Measured by threshold tracking nerve conduction studies

CONTACTS AND LOCATIONS:
Locations (1):
- Chiba University Hospital, Chiba, Japan